CLINICAL TRIAL: NCT04018742
Title: MICROBIOLOGY OF CEREBRAL ABSCESSES (ABCES)
Brief Title: MICROBIOLOGY OF CEREBRAL ABSCESSES
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-59; 2018-59 (Registry Identifier: APHM)
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Brain Abscess
MeSH Terms: conditions — Brain Abscess

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with an abscess: Patient diagnosed with a cerebral abscess at admission; and to benefit from an abscess puncture as part of routine care.
  Interventions: Other: Surgical puncture

INTERVENTIONS:
Other: Surgical puncture — Investigators propose to collect 20 abscesses. A collection of abscesses is performed systematically during the diagnostic for bacteriological analysis. There will be no further examination.

SUMMARY:
Establish the repertoire of bacteria and Archaea responsible for brain abscesses. Correlate the microbial repertoire to epidemiological, clinical and radiological data; to define the different nosological entities falling within the framework of cerebral abscesses.

DETAILED DESCRIPTION:
Brain abscess is a fatal infectious pathology of the central nervous system for which our CHU provides a referent function and supports patients suspected and diagnosed with a cerebral abscess in the area of the regional hospital group (GHT). Through the routine activity of the Microbiology laboratory of the IHU Méditerranée Infection, more than 180 diagnosed patients have been investigated in 9 years, an average of 20 patients per year. The mortality of brain abscesses is currently measured at 15% despite well-established diagnostic and therapeutic protocols in the literature, associating surgical drainage of abscess and administration of probabilistic antibiotics. Our hypothesis is that established protocols take into account incomplete microbiological documentation of cerebral abscesses and therefore anti-infectious therapy that may not be strictly adapted to the causative microorganisms. Our hypothesis is based on our own work as well as the literature data, showing that current approaches only target bacteria but that these approaches leave aside other living worlds such as Archaea. Indeed, investigators have recently shown for the first time that methanogens, which are Archaea microorganisms, constitute part of the flora responsible for certain cerebral abscesses and that they have a direct pathogenic role in cerebral abscesses. More specifically, the diagnosis of cerebral abscess includes several clinical and microbiological situations that are not all of the same therapeutic. Investigator propose to collect 20 abscesses. A collection of abscesses is performed systematically during the diagnosis for bacteriological analysis. There will be no further examination. The main objective of this clinical research project is to establish the repertoire of microorganisms responsible for brain abscesses; and as a secondary objective to define the different clinical entities forming the cerebral abscesses.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with a cerebral abscess at admission; and to benefit from an abscess puncture as part of routine care.
* Affiliate or beneficiary of a social security scheme.

Exclusion Criteria:

* Pregnant or nursing woman.
* Major patient under tutorship or curatorship.
* Patient deprived of liberty or under a court order
* Patient refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient diagnosed with a cerebral abscess at admission; and to benefit from an abscess puncture as part of routine care.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Matrix Assisted Laser Desorption Ionisation - Time of Flight | 1 day
  A matrix and a sample are deposited on a target. Pulsed lasers are fast charging.